CLINICAL TRIAL: NCT00208130
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Determine the Efficacy and Safety of Topiramate in the Treatment of Posttraumatic Stress Disorder in Civilians
Brief Title: Topiramate in the Treatment of Posttraumatic Stress Disorder in Civilians
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Frederick Petty, M.D., Creighton University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAPSS-201
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Topiramate

SUMMARY:
The primary objective of this study is to investigate the safety and efficacy of topiramate in the treatment of PTSD in women survivors of domestic violence and/or rape trauma as measured by the Clinician-Administered PTSD Scale (CAPS) for DSM-IV.

DETAILED DESCRIPTION:
Psychopharmacologic treatment of PTSD has been informed by only limited empirical data. Prior to the recently completed multi-site trials for sertraline conducted by Pearlstein and colleagues which found efficacy for women but not men suffering from chronic PTSD, there were only a handful of published randomized controlled trials. An overview of this literature suggests that tricyclic antidepressants, monoamine inhibitors and selective seratonin reuptake inhibitors (SSRIs) show promise, usually with better responses in civilians with PTSD than in male veterans with combat-related PTSD. Although results from open-label studies of alpha-2 agonists, beta blockers, anticonvulsants, and mood stabilizing agents appear to be promising, at present no one agent has emerged as useful for a broad range of PTSD sufferers.

This is a single-center, outpatient, randomized, double-blind, placebo-controlled, parallel group study designed to evaluate the safety and efficacy of topiramate in treating PTSD in civilian trauma. This study will be conducted in up to 60 subjects with a diagnosis of PTSD as defined by DSM-IV criteria. Thirty subjects will be assigned to topiramate and 30 will be assigned to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a diagnosis of PTSD as defined by DSM-IV for at least six months, supported by the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I).
2. Subjects must be female between 19 and 64 years of age, inclusive.
3. Subjects must have a minimum past week CAPS score of 50 at Visit 2 (Day 1).
4. Subjects must be in generally good health as confirmed by medical history, baseline psychiatric history and physical examination, including vital signs.
5. Subjects must have observed the designated washout periods for prohibited medications outlined under the Concomitant Therapy section of this protocol.
6. Subjects must have a negative urine drug screening (phencyclidine, cocaine, amphetamines, tetrahydrocannabinol, and opiates) at Visit 1.
7. Subjects must:

   1. be postmenopausal for at least one year, or
   2. have had a hysterectomy or tubal ligation or otherwise be incapable of pregnancy, or
   3. have practiced one of the following methods of contraception for at least one month prior to study entry: hormonal contraceptives, spermicide and barrier, intrauterine device, spousal/partner sterility or
   4. be practicing abstinence and agree to continue abstinence or to use an acceptable method of contraception (as listed above) should sexual activity commence.

   If (c) or (d), subjects must have a negative urine pregnancy test up to one week prior to Visit 2 (Day 1).
8. Subjects must be able to take oral medication, adhere to medication regimens and be willing to return for regular visits.
9. Subjects must be able to read and comprehend written instructions and willing to complete all scales and inventories required by this protocol.

Exclusion Criteria:

1. Subjects who have a DSM-IV diagnosis of substance dependence or abuse (with the exception of nicotine or caffeine dependence) within the past 3 months.
2. Subjects with a current or past history of primary major depressive disorder or major anxiety disorder (i.e., panic disorder, obsessive-compulsive disorder, social phobia) as defined by DSM-IV.
3. Subjects with a current or lifetime history of schizophrenia, bipolar disorder, or other psychotic disorder as defined by DSM-IV.
4. Subjects with a DSM-IV diagnosis of current organic mental disorder, factitious disorder, or malingering.
5. Subjects who are currently enrolled in a cognitive-behavioral therapy program.

   Note: Subjects may be receiving concurrent psychotherapy (other than cognitive-behavioral therapy), but subjects must not initiate new psychotherapy treatment during their participation in the trial.
6. Subjects with prior non-response to topiramate for the treatment of PTSD following an adequate trial.
7. Subjects with a disability or other compensation claim pending for lack of functioning due to PTSD.
8. Subjects with disability compensation dependent on persisting functional impairment related to PTSD.
9. Subjects who have previously been treated with topiramate and discontinued treatment due to an adverse event or subjects with a known hypersensitivity to topiramate.
10. Subjects with clinically unstable disease: cardiovascular, renal, gastrointestinal, pulmonary, metabolic, endocrine or other systemic disease that could interfere with their participation in the study.
11. Subjects with a history of nephrolithiasis.
12. Subjects who have SGOT and/or SGPT levels greater than 2 times the upper limit of the normal range at Screening.
13. Subjects who have active liver disease.
14. Subjects taking antipsychotics within three months of the screening visit.
15. Subjects with progressive or degenerative neurologic disorders (e.g., multiple sclerosis).

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60
Dates: Start 2001-10; Study Completion 2004-03

PRIMARY OUTCOMES:
The primary efficacy variable for this study will be the change of the 17-item total severity score of the CAPS from baseline to the last visit of Double-Blind Phase.

SECONDARY OUTCOMES:
The secondary efficacy variables consist of changes from baseline to the last visit in Double-Blind Phase of HARS, Ham-D, TOP-8 and CGI at the last visit of Double-Blind Phase.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Petty, MD, PhD, Principal Investigator — Creighton University
Locations (1):
- Creighton University Psychiatry and Research Center, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Monga V, Petty F, Padala K, Padala PR. Topiramate Monotherapy for Civilian Posttraumatic Stress Disorder: A Controlled Pilot Study. Prim Care Companion CNS Disord. 2023 Oct 19;25(5):23m03555. doi: 10.4088/PCC.23m03555. PMID 37857291